CLINICAL TRIAL: NCT03775499
Title: Proof of Concept Clinical Trial of Safety and Biological Activity of Bifidobacterium Longum NCC 2705 in Gluten Sensitivity
Brief Title: Probiotic BL NCC 2705 and Gluten Sensitivity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 17.11.NRC
Record Dates: First submitted 2018-11-01; First posted 2018-12-14 (Actual); Last update posted 2020-12-23 (Actual); Status verified 2020-12

CONDITIONS: Celiac Disease; Non-celiac Gluten Sensitivity
MeSH Terms: conditions — Celiac Disease | interventions — maltodextrin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Period 1: Placebo - Period 2: BL NCC 2705 (Other): For the 2 populations (Celiac and Non-Celiac Gluten Sensitivity)
  Interventions: Other: Intervention 1 : Maltodextrin; Dietary Supplement: Intervention 2 : BL NCC 2705 + Maltodextrin
- Period 1: BL NCC 2705 - Period 2: Placebo (Other): For the 2 populations (Celiac and Non-Celiac Gluten Sensitivity)
  Interventions: Dietary Supplement: Intervention 1 : BL NCC 2705 + Maltodextrin; Other: Intervention 2 : Maltodextrin

INTERVENTIONS:
Dietary Supplement: Intervention 1 : BL NCC 2705 + Maltodextrin — 2 capsules of BL NCC 2705/day (1 in the morning and 1 in the evening) for 3 days + 1 capsule of BL NCC 2705 in the morning of the 4th day
  Arms: Period 1: BL NCC 2705 - Period 2: Placebo
Other: Intervention 1 : Maltodextrin — 2 capsules of Placebo/day (1 in the morning and 1 in the evening) for 3 days + 1 capsule of Placebo in the morning of the 4th day
  Arms: Period 1: Placebo - Period 2: BL NCC 2705
Dietary Supplement: Intervention 2 : BL NCC 2705 + Maltodextrin — 2 capsules of BL NCC 2705/day (1 in the morning and 1 in the evening) for 3 days + 1 capsule of BL NCC 2705 in the morning of the 4th day
  Arms: Period 1: Placebo - Period 2: BL NCC 2705
Other: Intervention 2 : Maltodextrin — 2 capsules of Placebo/day (1 in the morning and 1 in the evening) for 3 days + 1 capsule of Placebo in the morning of the 4th day
  Arms: Period 1: BL NCC 2705 - Period 2: Placebo

SUMMARY:
The aim of the study is to confirm/prove safety of the probiotic and production of serpin in humans.

DETAILED DESCRIPTION:
This trial is a multicenter, double blind, randomized, placebo controlled, 2 by 2 cross-over design (i.e. 2-sequences, 2-periods, 2-treatments) for each specific population (i.e. self-reported Non Coeliac Gluten Sensitivity and Coeliac Disease subjects).

1 capsule of BL NCC 2705 or placebo will be given twice a day in the morning and in the evening with a meal over 2 periods of 4 days.

On day four a single dose of gluten (3g) will be administered and duodenal fluid will be collected in the following hours through a naso-intestinal catheter. The viability of BL NCC 2705, the production of serpin and its effects on gluten digestion and intestinal enzymatic activity will be determined.

No chronic administration of gluten as a challenge is foreseen in the study.

After a wash out period of minimum 2 weeks, period will be repeated.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to sign written informed consent prior to trial entry
2. Male or female adults >18 years of age
3. For NCGS: self-reported gluten sensitivity with negative CD serology, on gluten free diet for at least 6 weeks with self-reported significant symptomatic improvement
4. For CD: confirmed serologic and histologic diagnosis of CD and on GFD for at least 12 months with self-reported significant symptomatic improvement
5. Body Mass Index (BMI) within the range >18 - <30 kg/m2
6. Willing and able to comply with study procedures and restrictions
7. In good health as determined by a medical history and medical examination

Exclusion Criteria:

1. Documented IgE-mediated food allergy
2. Subjects following an overly imbalanced or restrictive diet as per nutritional advice
3. Concurrent systemic disease and/or laboratory abnormalities considered by investigators to be detrimental for the participants safety or potentially interfering with the study procedures and/or study outcomes
4. Concurrent organic GI pathology other than benign polyps, diverticulosis, hemorrhoids, lipomas and melanosis coli
5. Previous abdominal surgery with the exception of hernia repair, appendectomy, caesarian section, tubal ligation, hysterectomy, hemorrhoidectomy
6. Patients who received antibiotics in the previous 2 weeks
7. women of childbearing potential not willing to use an effective contraception method

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2018-10-09 (Actual); Primary Completion 2019-10-04 (Actual); Study Completion 2020-12-15 (Actual)

PRIMARY OUTCOMES:
incidence, type and severity of adverse event | from Baseline to end of study (up to maximum 43 days)
  incidence, type and severity of adverse event
Gastro-intestinal tolerability: visual analog scale | from Baseline to end of study (up to maximum 43 days)
  Sum of visual analog scale for gastro-intestinal symptoms assessment (nausea, vomiting, diarrhea, audible bowel sound, flatulence and abdominal cramping symptoms are assessed). Each scale is from 0 (no symptom) to 100mm (maximum symptom). The maximum sum value is 600.

SECONDARY OUTCOMES:
Concentration of bacterial Serpin RNA and/or proteins (ng/mL) in duodenal aspirates | 19 sampling over 6h50 hours at visit 2 (day 4) and visit 3 (from day 22 to day 36)
  Measurements via RT-PRC and immuno-assay
Concentration of Probiotic BL NCC 2705 (ng/mL) in duodenal aspirates | 19 sampling over 6h50 hours at visit 2 (day 4) and visit 3 (from day 22 to day 36)
  Measurements via PCR
Concentration of gluten derived pepides in duodenal aspirates | 10 sampling over 3h30 at visit 2 (day 4) and visit 3 (from day 22 to day 36)
  Effect of BL NCC 2705 on gluten digestion based on the amount of gluten peptides detected in duodenal apsirates
Concentration of gluten derived pepides in urine | 10 sampling over 3h30 at visit 2 (day 4) and visit 3 (from day 22 to day 36)
  Effect of BL NCC 2705 on gluten digestion based on the amount of gluten peptides detected in urine
Level of elastase (Units/ mL) activity in duodenal aspirates | 19 sampling over 6h50 hours at visit 2 (day 4) and visit 3 (from day 22 to day 36)
  Measurements of proteolytic activity based assay

CONTACTS AND LOCATIONS:
Overall Officials: Carmine D'Urzo, Dr., Study Director — Nestec Ltd.
Locations (1):
- Viecuri Hospital, Venlo, Netherlands